CLINICAL TRIAL: NCT01552174
Title: Management of Eyelid Disorders by Ophthalmologists in Usual Medical Practice
Acronym: MEIBUM
Status: Completed | Type: Observational
Sponsor: Laboratoires Thea (Industry)
Collaborators: Iris Pharma (Industry); Axial Biotech, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: MEIBUM survey
Record Dates: First submitted 2012-03-06; First posted 2012-03-13 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Palpebral Pathologies; Ocular Surface Disease; Meibomian Gland Dysfunction
Keywords: MGD; ocular surface pathologies
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Outpatients attending general ophthalmologic consultation: * Outpatients of either sex, aged at least 18 years, seen in general ophthalmological consultation
  * Patients informed of the objectives of the survey and agreeing to participate.
  * Patient attending to the ophthalmological consultation for any reasons: regular check-up of chronic disease, acute symptoms, or for surgery preparation or follow up.

SUMMARY:
The purpose of this study is to determine the incidence and characteristics of eyelid inflammatory disorders during general ophthalmological consultations and to demonstrate association between palpebral pathologies and ocular surface pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients of either sex, aged at least 18 years, seen in general ophthalmological consultation
* Patients informed of the objectives of the survey and agreeing to participate.
* Patient attending to the ophthalmological consultation for any reasons: regular check-up of chronic disease, acute symptoms, or for surgery preparation or follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be eligible for inclusion if all these criteria are respected:
  * Outpatients of either sex, aged at least 18 years, seen in general ophthalmological consultation
  * Patients informed of the objectives of the survey and agreeing to participate.
  * Patient attending to the ophthalmological consultation for any reasons: regular check-up of chronic disease, acute symptoms, or for surgery preparation or follow up.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Incidence of eyelid disorders in general ophthalmological practice | Day 1
  * Systematic description of the eyelid, the ocular surface and the dermatological aspect of the face
  * Occurrence of Meibomian Gland Dysfunction(MGD).

SECONDARY OUTCOMES:
Association between palpebral pathologies and ocular surface pathologies | Day 1
  To describe association between palpebral pathologies and ocular surface pathologies
Impact of eyelid disorder on patient's daily life | Day 1
  Consequences on vision, on daily life activities/work, on leisure, on contact lens wearing, on emotions, on sleeping,
Current recommended strategy to treat eyelids disorders | Day 1
  Description of recommended strategy

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel Benitez del Castillo, Professor, Principal Investigator — USIO, Departamento de Oftalmología, Hospital Clínico San Carlos, 28040 Madrid, Spain
Locations (2):
- Consultation office, Heidelberg, Germany
- USIO Departamento de Oftalmologia Hospital Clínico San Carlos, Madrid, Spain